CLINICAL TRIAL: NCT01304927
Title: Vitamin D Supplementation and Male Infertility: The Copenhagen Bone-Gonadal Study a Double Blinded Randomized Clinical Trial
Brief Title: Vitamin D Supplementation and Male Infertility: The CBG-study a Randomized Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin Blomberg Jensen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010124801; 2010-024588-42 (EudraCT Number); H-4-2010-138 (Other: Ethical committee)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Male Infertility
Keywords: Reproduction; Sex hormones; Glucose metabolism; Bone metabolism; Calcium; Sperm; testis; bone; endocrinology
MeSH Terms: conditions — Infertility, Male | interventions — Cholecalciferol; Calcium; Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol + calcium (Active Comparator): Group of intervention: Each man will receive 300,000 IU (7500 ug) Cholecalciferol (VD3) orally once after blood and semen sampling and performed DXA scan. Thereafter they will receive VD tablets of 1,400 IU (35 ug) + 500 mg calcium daily for 3 months. At 3 months a clinical control and blood sampling will be performed, followed by continued daily intake of 1400 IU VD3 + 500 mg calcium. At end of treatment at five months after inclusion the men deliver two semen samples, have a blood sample drawn and a DEXA scan performed.
  Interventions: Drug: Cholecalciferol and calcium
- placebo (Placebo Comparator): Group receiving placebo: Each man will receive placebo oral mixture once after blood- and semen sampling and performed DXA scan. Thereafter they will receive placebo tablets daily for 3 months. At 3 months a clinical control and blood sampling will be performed, followed by continued daily intake of placebo. At end of treatment at five months after inclusion the men deliver two semen samples, have a blood sample drawn and a DEXA scan performed.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol and calcium — Initial one dose oral mixture of 300.000 IU Cholecalciferol followed by 5 months treatment with one tablet daily containing 35 ug Cholecalciferol and 500 mg calcium
  Other Names: Inactive vitamin D
  Arms: Cholecalciferol + calcium
Other: Placebo — microcrystalline cellulose maltodextrin Arachidis oil
  Arms: placebo

SUMMARY:
Today, it is evident that vitamin D (VD) has more widespread effects than the classical actions related to bone mineralization and calcium homeostasis1. VD deficiency results in impaired reproductive performance in various species of animals, and recently the investigators have shown that the VD receptor (VDR), activating (CYP2R1, CYP27A1, CYP27B1) and inactivating (CYP24A1) enzymes are expressed in the human testis, epididymis, seminal vesicle, prostate and spermatozoa. Our following functional studies showed that VD increases intracellular calcium in mature spermatozoa, and hence may be important not only for spermatogenesis but also for sperm maturation. A new, and yet unpublished cross sectional study of 300 young healthy Danish men showed that men with lower levels of serum VD have significantly lower number of normally developed and motile spermatozoa. Hitherto, most cases of male infertility have been classified as "idiopathic", and infertile couples have been referred to symptomatic treatment at infertility clinics. These fertility treatments are often physically demanding for the female partner as well as expensive for the health care system. Any treatment that might improve semen quality of involuntary infertile men would be beneficial both for the infertile couples and the society in general. Our findings that VD may play a role for human semen quality have not yet been tested clinically. However, if VD supplementation proves efficient this opens for the first time for a causal, safe and cheap treatment of at least some cases of "idiopathic" impaired semen quality. The investigators believe our new human data supported by the results from the VD deficient and VDR KO animal studies and the high proportion of VD deficient Danish men provide sufficient evidence to initiate a randomized clinical trial of VD supplementation to infertile men. Infertile men have also have unfavorable altered levels of sex hormones and higher mortality than fertile men. Since VD deficiency is associated with increased mortality, regulation of aromatase, immune system, bone metabolism, glucose metabolism, cardiovascular system etc. our suggested clinical trial may also be able to evaluate several secondary endpoints in addition to the potential effect on semen quality.

DETAILED DESCRIPTION:
Background In 2008, approximately 8% of all newborn children were conceived by assisted reproduction. Intracytoplasmatic sperm injection (ICSI) accounts for ~50% of all treatments and is mainly used in cases of severely reduced semen quality. This is in many cases most likely caused by prenatal factors adversely affecting the developing testicles, and it is therefore unlikely that any treatment of adult men will be able to completely normalize their semen quality. However, less would also be clinically relevant. If reduced semen quality could be improved prior to any assisted reproduction a less invasive treatment would be needed. Eg. classical in vitro fertilization (IVF) rather than ICSI, simple intrauterine insemination (IUI) rather than IVF or natural conception rather than IUI.

Several endocrine factors have been implicated in sperm production and maturation, but little is known about the potential role of VD. VD is a key regulator of calcium homeostasis and bone mineralization, although expression of the vitamin D receptor (VDR) in various tissues has been related to several diverse actions. VD affects reproduction in several animal species, convincingly shown in rodents, where VD deficiency in male rats resulted in reduced sperm counts, and female rats inseminated with semen from VD deficient male rats had lower fertility rates. The impaired reproductive performance is reversible and can be corrected either by supplying VD or by normalizing calcium levels. Supported by VDR knockout mice, which showed decreased sperm counts, reduced sperm motility and histological abnormalities of the testis, which unlike the VD deficient male rats only partly can be restored by calcium supplements.

The investigators have recently shown expression of VDR and the VD metabolizing enzymes in the human testis, ejaculatory tract and in mature spermatozoa. The investigators subsequently showed that VD in physiological concentrations increased intracellular calcium in spermatozoa. VD acts through a rapid non-genomic response and the VD induced increase in calcium may be crucial for the spermatozoa, because VD induced sperm motility and the acrosome reaction. Expression analysis of spermatozoa from fertile and infertile men showed that men with impaired semen quality have fewer that can metabolize VD than normal men(p < 0.0005) making presence of one of the proteins a potential marker of semen quality. Furthermore, the investigators have just completed a cross sectional study of 300 young men from the general population and found that low serum VD was associated with reduced sperm motility and morphology.

SETTING, SCIENTIFIC PLAN AND RECRUITMENT Participants will be included among men referred to the Department of Growth and Reproduction (dept. of GR), Rigshospitalet (RH) for evaluation of male infertility

DESIGN This is a prospective, double blinded, two-arm randomized controlled trial

Group of intervention: Each man will receive 300,000 IU (7500 ug) cholecalciferol (D3) orally once after blood- and semen sampling and performed DXA scan. Thereafter they will receive VD tablets of 1,400 IU (35 ug) + 500 mg calcium daily for 3 months. Telephone control after 4 weeks and at 3 months a clinical control and blood sampling will be performed, followed by continued daily intake of 1400 IU VD + 500 mg calcium for 2 additional months. At end of treatment at five months after inclusion the men deliver two semen samples, have a blood sample drawn and a DXA scan performed.

Group receiving placebo: Will follow the same chain of events, although VD will be replaced with placebo.

PARTICIPANTS Screening of ~700-800 infertile men will be performed. The investigators assume that ~340 men will be excluded and ~100 men do not wish to participate. Thus, 300 men will be included in the study and half will be randomized to active VD treatment. The investigators expect a small drop out (< 20) because of high motivation and no adverse effects.

ANALYSIS AND INTERVENTION Reproductive hormones and growth factors will be analyzed at dept. of GR, Rigshospitalet. An aliquot of the first blood sample will be analyzed before inclusion to the study and another kept to be analyzed at the same time as the second blood sample at the end of the trial to overcome the interassay variation. Other serum analyses will be analyzed at department of clinical biochemistry, Rigshospitalet. Semen analyses and DXA scans will be performed at dept. of GR.

SAMPLE SIZE CALCULATION AND STATISTICS In our association study with 300 participants the investigators are able to detect significant dose response relationship between VD status and sperm motility and morphology, and found significant differences between men with low and high VD levels. Based on these results, the investigators assume to be able to increase serum levels of VD with 50 nM with our setup. Including 150 men in each group will enable us to detect changes in sperm motility and morphology of 15% and a 25% change in Inhibin B levels. Intention to treat principles will be used and co-variate analyzes will be used to analyze the potential effect of VD.

BIOSTATISTICAL ANALYSIS All the analyses will be performed according to Good Clinical Practice guidelines and the primary analyses in the intention-to-treat population, which included all patients who underwent randomization and received the first dose of medicine on day 1. We will analyze the data in 3 ways. The primary analysis will proceed according to the randomized vitamin D and calcium dose group assignment. The secondary analysis will be based on stratifying the men according to subgroup analyses in relation to the predefined primary and secondary endpoints, while the last analysis will try to elucidate any dose-response relationship. An author (JHP) who was the statistician for the study and unaware of the study-group assignments will perform the primary analysis.

Data analysis and quality The primary end points for this protocol will be changes in semen quality especially sperm motility followed by sperm concentration, morphology and semen volume. Multiple secondary endpoints exist but for the initial investigation focus will be on changes of the following secondary endpoints: Sperm DFI, pregnancy rate, Inhibin B, vitamin D and calcium homeostasis. Subjects who terminate participation after visit at 90 days but before visit day 150 will be included for data analysis up to day 90. Men that only deliver one semen sample or have missing data at any visit will still be included in the analysis. Men with fever up to 3 months prior to semen analysis will be considered as a potential confounder. Men that do not meet the criteria in the protocol will be excluded from the analysis. Those values will then be carried forward for analyses. A significance level of 5% is used. For the primary analyses Bonferronu-Holm p-value correction is calculated additionally. For the secondary analysis no multiple test correction are used. Instead results are discussed in view of the multiple testing situations.

1. Analyses between placebo versus active substance Between group analyses placebo versus vitamin D + calcium: The first step will be to compare the changes in primary outcomes across the two groups placebo versus vitamin D + calcium. This analysis will show if there is a significant difference between groups. For outcomes measured repeatedly, this will entail comparing the estimated slopes, or rates of change, of each outcome between the groups. Mixed models allow for the correlation between the repeated observations baseline-day 1-day 90- day 150 from each man to be suitably incorporated into parameter estimation. For all endpoints measured at baseline and day 150, paired t-tests will be used to assess there is a significant difference between the groups and determine whether the mean change within each group differs significantly from zero. In both cases, data will be transformed as necessary to meet model assumptions. Afterwards, the same analysis will be conducted by using multiple regression with relevant confounders such as season, BMI, smoking, duration of abstinence, time from ejaculation to motility assessment, fever etc. to see if this changes the results For outcomes measured that cannot be compared with t-test or other parametric tests at day 1, day 90 and day 150, groups will be compared using non-parametric tests such as Wilcoxon Mann-Whitney test. For Binary outcome the data will be compared between the two groups by means of conditional logistic-regression analysis with adjustment for relevant confounders (defined as being significantly p<0.05 associated).

   .
2. Analyses after stratification into subgroups Subjects will be grouped according to their BMI, calcium, season, semen quality, bonefactors, BMD or vitamin D levels and the effect of placebo versus active substance will be evaluated at day 90 and day 150. The subgroup analyses will in accordance with normal clinical practice and stratification in appropriate groups according to the clinical (25OHD < 25 nmol/l, BMI <25, 25-30, >30 etc.), tertiles/quartiles/quintiles or highest/lowest versus remaining at baseline.
3. Data analysis for comparison of changes in vitamin D and calcium We will also compare the dose-response relationships between changes in vitamin D and calcium and primary and secondary endpoints between placebo and active substance group and in all men. We will determine delta values for circulating vitamin D progenitors, calcium ion, total calcium and albumin corrected calcium from start to 90 days and 150 days and compare the difference with the observed changes in primary and secondary endpoints. We anticipate that there is no difference in shapes of the dose-response curve between the different endpoints i.e. they will be parallel and linear at least after transformation of the data. Afterwards, the same analysis will be conducted by using relevant confounders such as season, BMI, smoking, duration of abstinence, time from ejaculation to motility assessment etc. to see if this changes the results.

SCREENING AND TIME COURSE Men, who are investigated at dept. of GR due to infertility will be screened for eligibility to the study, and those who meet the criteria for participation will be informed, and if they consent allocated to active treatment with VD or placebo. Allocation will be done by minimization using minim to avoid unbalanced grouping due to randomization failure. Following variables will be balanced: Sperm concentration, BMI, serum inhibin-B, and VD level.

ETHICS AND SIDE EFFECTS All the patients will have fulfilled their investigation, before they are invited to the study. They will be informed of potential adverse effects, signs of intoxication and they can leave the trial at any point without any consequences. The trial will run in accordance with "good clinical practice". VD treatment gives virtually no side effects and the risk of intoxication is almost nonexisting in the suggested setting, with relatively low doses of VD and close monitoring of VD and calcium status. The participants will be exposed to oral VC/placebo, to 2 DXA scans, have 3 extra blood samples drawn and deliver 2 extra semen samples. All participants will be informed and counseling according to their VD status.

PUBLICATION OF RESULTS All results, positive or negative will be submitted to peer reviewed scientific journals. Data will successively be obtained and transferred to a statistical database.

PRACTICAL ISSUES Dept. of GR investigates annually more than 500 infertile men. Participants will be included from that group. The department have the clinical expertise, experience and capacity to perform all the investigations, except for the measurements of some of the blood samples, which will be analyzed by department of clinical biochemistry. VD and placebo oral suspensions are purchased from Glostrup apotek, while VD and placebo tablets are purchased from Ferrosan, MD Martin. The investigators are collaborating with associate professor in biostatistics J.H. Petersen, University of Copenhagen.

ELIGIBILITY:
Inclusion Criteria:

* Male with an age > 18 years old
* Referred for male infertility with sperm concentration >= 0.01 million/ml. Additionally, all men must have either sperm concentration < 20 million/ml or < 50% progressive motile spermatozoa or < 12% morphological normal spermatozoa using strict criteria

Exclusion Criteria:

* Men with chronic diseases (such as diabetes mellitus, Thyroid disease, endocrine disturbances in need of treatment, malignant disease, or diseases known to interfere with VD intake or very sensitive to VD intake (such as inflammatory disease with granuloma: sarcoidoses, tuberculosis, Wegeners, vasculitis, inflammatory bowel disease (Crohn's and colitis ulcerosa etc).
* Men with present or previous malignant disease
* If there is an indication for testis biopsy and it is planned or conducted within the next 6 months
* Serum 25-hydroxy-D3 > 50 nmol/l at the time of inclusion
* Serum Calcium ion > 1,35 mmol/l
* Inhibin-B < 30 pg/ml
* Intake of vitamin D above 15 ug daily
* Allergy towards vitamin D or arachidis oil (peanuts)
* Men with total or partly obstructive oligospermia and men who had vasectomy performed

Criteria for drop out:

* Abrogation of the treatment
* Newly diagnosed endocrine, calcium metabolic disease, parathyroid, thyroid, diabetes or other endocrine disease in need of treatment
* New malignant disease
* Treatment with chemotherapy, immunomodulating therapy, salazopyrin
* Oral or iv treatment with steroid hormones
* Treatment with diuretics, antihypertensive treatment, treatment the heart, calcium channel blockers
* Development of vitamin d intoxication
* If testis biopsy is performed or other surgery in the genital region during the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
semen quality | 150 days
  difference in semen quality (semen variables total sperm count, sperm concentration, sperm motility, sperm morphology and semen volume) between VD and placebo treated men after 150 days of treatment.
sperm motility | 150 days
  Differences in Sperm motility (ABC) and progressive sperm motility (AB) between placebo and VD group, supported by other motility measures such as length of penetration in egg media and difference in motility over time (3-5 hours from ejaculation)between VD and placebo treated men
sperm morphology | 150 days
  Differences in percentage of spermatozoa with normal morphology assessed according to strict criteria between placebo and VD group.
sperm concentration | 150 days
  Differences in sperm concentration between placebo and VD group.
total sperm count | 150 days
  Differences in total sperm count between placebo and VD group.
semen volume | 150 days
  Differences in semen volume between placebo and VD group.

SECONDARY OUTCOMES:
Inhibin-B | 90 and 150 days
  Difference in serum levels of Inhibin B between placebo and VD group after 90 and/or 150 days
Testosterone | 90 and 150 days
  Difference in serum levels of total and free testosterone between placebo and VD group after 90 and/or 150 days
AMH | 90 and 150
  Difference in serum levels of anti-müellerian hormone (AMH) between placebo and VD group after 90 and/or 150 days
estrogen | 90 and 150
  Difference in serum levels of estrogen (estradiol) between placebo and VD group after 90 and/or 150 days
LH | 90 and 150 days
  Difference in serum levels of lh (luteinizing hormone) between placebo and VD group after 90 and/or 150 days
FSH | 90 and 150 days
  difference in FSH (follicle stimulating hormone) between placebo and VD group after 90 and/or 150 days
SHBG | 90 and 150 days
  difference in SHBG (sex hormone binding hormone) between placebo and VD group after 90 and/or 150 days
DXA scan | 150 days
  difference in fat mass, fat free mass, muscle mass and bone mineral density evaluated by full body DXA scan between placebo and VD group after 150 days
Circulating metabolites of Vitamin D | 90 and 150 days
  difference in the following VD metabolites inactive VD2 and VD3,25-hydroxy-VD2, 25-hydroxy-VD3, 1,25(OH)2D3, 24,25(OH)2D3, and 1,24,25(OH)2D3 between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
PTH | 90 and 150 days
  difference in the following serum levels of PTH (parathyroid hormone between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
alkaline phosphatase | 90 and 150 days
  difference in the following serum levels of alkaline phosphatase (also bone specific subtype) between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
calcium | 90 and 150 days
  difference in the following serum levels of calcium ( meaning total calcium, calcium ion and albumin corrected calcium) between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
phosphate | 90 and 150 days
  difference in the following serum levels of phosphate between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
FGF23 | 90 and 150 days
  difference in the following serum levels of FGF23 (both intact and fragmented) between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
Klotho | 90 and 150 days
  difference in the following serum levels of klotho (also subtypes) between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
osteocalcin | 90 and 150 days
  difference in the following serum levels of osteocalcin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
osteopontin | 90 and 150 days
  difference in the following serum levels of osteopontin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
Rank-L | 90 and 150 days
  difference in the following serum levels of Rank-L between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
calcitonin | 90 and 150 days
  difference in the following serum levels of calcitonin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
bone markers | 90 and 150 days
  difference in the following serum levels of bone markers such as procollagen III between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
change in the method of assisted reproductive technique or number of pregnancies | 90 and 150 days
  difference in the type of method used IUI, IVF, ICSI and in the number of achieved pregnancies between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
change in the number of spontaneous pregnancies | 90 and 150 days
  difference in the number of spontaneous achieved pregnancies between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
blood pressure | 90 and 150 days
  difference in systolic and/or diastolic blood pressure between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
CYP24A1 expression at the annulus | 150 days
  difference CYP24A1 expression at the annulus of human spermatozoa between placebo and VD group after 150 days and between the initial level (day 0) and 150 days in both arms.
Bone and calcium regulators in seminal fluid | 150 days
  difference in seminal fluid concentration of pH, HCO3-, calcium, zinc, phosphate, VD, 1,25(OH)2D3, 25-OHD3, 24,25(OH)2D3, 1,24,25(OH)2D3, FGF23, Klotho, osteocalcin, osteopontin between placebo and VD group after 150 days and between the initial level (day 0) and 150 days in both arms.
weight and BMI | 90 and 150 days
  difference in weight and BMI between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
Glucose metabolism | 90 and 150 days
  difference in serum level of glucose, Hb1Ac, cholesterol, lipid profile, insulin, leptin, adiponectin, C-peptid, HOMA, insulin sensitivity, incretin hormones (such as GLP1 and 2)between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
Growth and IGF axis | 90 and 150 days
  difference in serum level of GH, IGF-I, IGFBP-3 between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
tumor markers | 90 and 150 days
  difference in PSA (prostate specific antigen both free and bound) and CEA ( carcino embryonic antigen)between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
stress hormones | 90 and 150 days
  difference in serum level of cortisol, ACTH and copeptin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
prolactin | 90 and 150 days
  difference in serum level of prolactin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
kidney and cardiovascular markers | 90 and 150 days
  difference in serum level of creatinin, albumin, urea, urea acid (urat), creatinine clearance, renin, aldosteron, angiotensinogen, B2-microglobulin, and angiotensin 2 between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
liver markers | 90 and 150 days
  difference in serum level of aminotransferases (ALAT, ASAT, GGT), LDH, amylase, bilirubin between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
infectious disease | 28, 90 and 150 days
  difference in frequency and severity of infectious diseases such as cold, sinusitis, tonsillitis, laryngitis, pneumonia, UVI, gastroenteritis, skin infections. between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
fever | 28, 90 and 150 days
  difference in frequency and severity of fever episodes between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
inflammatory markers | 90 and 150 days
  difference in the following serum levels of acute phase reactants such as CRP (C reactive peptide), Ferritin, procalcitonin, leukocytes, thrombocytes, reticulocytes, RBC, haematocrit, complement, immunoglobulins, auto-antibodies such as ANA, antiphopholipantibody, rheumafactor and coagulation factors between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
natriuretic peptides | 90 and 150 days
  difference in the following serum levels of ANP and BNP between placebo and VD group after 90 and/or 150 days and between the initial level (day 0) and 90 and 150 days in both arms.
DNA Fragmentation | 0-150
  DNA fragmentation index will be investigated on 75-100 randomly selected individuals prior to and following the intervention with either placebo or vitamin D
Predefined Subgroup analyses | day 90 and 150
  Predefined subgroups. Vitamin D levels: a. deficient< 25 nM, b. insufficient 25-50 nM Season: a. Winter, b. spring, c. summer and d. autumn or x. Winter(October-March)and y.Summer(April to September) Serum calcium ion: a. =/<1.20 nM , b. > 1.20 nM Sperm concentration: a. < 5 million/ml, b. 5-20 million/ml,c. > 20 million/ml Inhibin B: a. < 100 pg/ml ,b. 100-150 pg/ml, c. > 150 pg/ml BMI: a. < 25 , b. 25-30, c. > 30 Cryptorchidism: a. YES/NO

CONTACTS AND LOCATIONS:
Overall Officials: Martin Blomberg Jensen, MD, Principal Investigator — Department of growth and reproduction, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Yahyavi SK, Toft FB, Probst-Drejer B, Boisen IM, Priskorn L, Jorgensen N, Juul A, Blomberg Jensen M. High Seminal Fluid Calcium Is Associated With Higher Sperm Concentration in Infertile Men and Men From the General Population. Andrology. 2026 Jan 14:e70172. doi: 10.1111/andr.70172. Online ahead of print. PMID 41531256
- [Derived] Wall-Gremstrup G, Holt R, Yahyavi SK, Jorsal MJ, Juul A, Jorgensen N, Blomberg Jensen M. High-dose vitamin D3 supplementation shows no beneficial effects on white blood cell counts, acute phase reactants, or frequency of respiratory infections. Respir Res. 2024 Jan 4;25(1):11. doi: 10.1186/s12931-023-02642-9. PMID 38178229
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389
- [Derived] Holt R, Petersen JH, Dinsdale E, Knop FK, Juul A, Jorgensen N, Blomberg Jensen M. Vitamin D Supplementation Improves Fasting Insulin Levels and HDL Cholesterol in Infertile Men. J Clin Endocrinol Metab. 2022 Jan 1;107(1):98-108. doi: 10.1210/clinem/dgab667. PMID 34508607
- [Derived] Juel Mortensen L, Lorenzen M, Jorgensen A, Albrethsen J, Jorgensen N, Moller S, Andersson AM, Juul A, Blomberg Jensen M. Possible Relevance of Soluble Luteinizing Hormone Receptor during Development and Adulthood in Boys and Men. Cancers (Basel). 2021 Mar 16;13(6):1329. doi: 10.3390/cancers13061329. PMID 33809538
- [Derived] Juel Mortensen L, Lorenzen M, Jorgensen N, Andersson AM, Nielsen JE, Petersen LI, Lanske B, Juul A, Hansen JB, Blomberg Jensen M. Possible link between FSH and RANKL release from adipocytes in men with impaired gonadal function including Klinefelter syndrome. Bone. 2019 Jun;123:103-114. doi: 10.1016/j.bone.2019.03.022. Epub 2019 Mar 23. PMID 30914274
- [Derived] Blomberg Jensen M, Lawaetz JG, Petersen JH, Juul A, Jorgensen N. Effects of Vitamin D Supplementation on Semen Quality, Reproductive Hormones, and Live Birth Rate: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Mar 1;103(3):870-881. doi: 10.1210/jc.2017-01656. PMID 29126319
- [Derived] Blomberg Jensen M, Gerner Lawaetz J, Andersson AM, Petersen JH, Nordkap L, Bang AK, Ekbom P, Joensen UN, Praetorius L, Lundstrom P, Boujida VH, Lanske B, Juul A, Jorgensen N. Vitamin D deficiency and low ionized calcium are linked with semen quality and sex steroid levels in infertile men. Hum Reprod. 2016 Aug;31(8):1875-85. doi: 10.1093/humrep/dew152. Epub 2016 Jun 19. PMID 27496946